CLINICAL TRIAL: NCT04106115
Title: A Phase Ib/II Study to Assess the Safety and Activity of DURvalumab (MEDI4736) in Combination With S-488210/S-488211 vAccine in Non-muscle Invasive Bladder CancEr
Brief Title: DURvalumab in Combination With S-488210/S-488211 vAccine in Non-muscle Invasive Bladder CancEr
Acronym: DURANCE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry); Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/121881
Record Dates: First submitted 2019-09-09; First posted 2019-09-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer
Keywords: Non-Muscle Invasive Bladder Cancer (NMIBC); Durvalumab; S-488210/S-488211; Immunotherapy; Vaccine; PD-L1 Inhibitor; BCG unresponsive
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — durvalumab; Monatide (IMS 3015)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + S-488210/S-488211 (Experimental): Trial treatment for up to 24 weeks of Durvalumab (1500 mg IV infusion every 4 weeks for up to 7 doses) in combination with S-488210/S-488211 vaccine (given as 2 subcutaneous injections of S-488210/Montanide and S-488211/Montanide starting day after first durvalumab dose, then weekly for the first 6 weeks, and then every 2 weeks for a further 9 doses).
  Interventions: Drug: Durvalumab; Biological: S-488210/S-488211

INTERVENTIONS:
Drug: Durvalumab — 1500 mg IV infusion every 4 weeks for up to 7 doses
  Other Names: MEDI 4736
Biological: S-488210/S-488211 — S-488210/S-488211 is given as a 1 mL subcutaneous (SC) injection of S-488210/Montanide emulsion and a 1 mL SC injection of S-488211/Montanide emulsion starting the day after first dose of durvalumab and continuing weekly for 6 doses and then every 2 weeks for a further 9 doses
  Other Names: S-488210/Montanide; S-488211/Montanide

SUMMARY:
DURANCE is a two part, phase Ib/II, multi-centre study to assess the safety and activity of S-488210/S-488211 in combination with durvalumab, in patients with non-muscle invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
DURANCE is a registered, phase Ib/II study in patients with surgically debulked bacillus Calmette-Guerin (BCG) unresponsive (resistant or relapsing) or intolerant non-muscle invasive bladder cancer (NIMBC). Patients will receive up to 24 weeks of durvalumab (a PD-L1 immune checkpoint inhibitor) in combination with S-488210/S-488211 (a 5-peptide cancer vaccine).

Durvalumab will be given as 1500 mg IV infusion every 4 weeks for up to 7 doses, in combination with S-488210/S-S488211 which will be administered as two subcutaneous injections of S-488210/Montanide and S-488211/Montanide starting the day after the first durvalumab dose, then weekly for 6 doses and every 2 weeks for a further 9 doses (up to a maximum of 16 doses).

All patients must have a cystoscopy at the end of week 12 (from start of trial treatment) for disease evaluation and to assess suitability to continue trial treatment. Patients with complete response, as shown from the cystoscopy, may continue treatment for up to 24 weeks in the absence of progressive disease, unacceptable toxicity or withdrawal of consent; all other patient will be withdrawn from further trial treatment.

The phase Ib part of the DURANCE study will look to assess the safety and tolerability of the treatment combination of durvalumab + S-488210/S-488211 by reviewing Dose Limiting Toxicities (DLTs) which have at least a reasonable possibility of being related to the trial treatments (durvalumab and/or S-488210/S-488211). Up to 14 evaluable patients will be registered into phase Ib and provided the DLTs do not exceed the DLT thresholds defined in the trial protocol, the trial will proceed to the expansion phase of the study (phase 2). In phase 2 the trial will look to assess the disease free survival rate at 1 year following start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven high risk non-muscle invasive bladder cancer (NMIBC)
2. Adequate archival tissue sample available for histological assessment (date sample taken must be within 6 months of planned start of treatment)
3. Predominant histologic component (> 50%) must be urothelial (transitional cell) carcinoma
4. Bacillus Calmette-Guerin (BCG) unresponsive disease or are intolerant of BCG therapy
5. Refused or deemed clinically inappropriate for radical cystectomy
6. ≥18 years of age
7. Body weight >30 kg
8. World Health Organisation (WHO) performance status 0-1
9. Must have undergone each of the following procedures within 8 weeks of registration:

   * Complete excision of all papillary disease (T1/TaHG) and demonstration of no muscle invasive disease in the resected specimens (muscle must be present in the tumour sample)
   * Bladder 'Mapping biopsies' taken
   * CT of the chest
   * CT Urogram or MRI of the abdomen and pelvis (if CT is not possible)
10. Adequate haematological status:

    * Haemoglobin ≥9.0 g/dL
    * Absolute neutrophil count ≥1.5 x 10^9/L (≥150,000 per mm3)
    * Platelet count ≥100 x 10^9/L (≥100,000 per mm3)
    * International Normalised Ratio (INR) ≤1.5 and Activated Partial Thromoplastin Time (APTT) ≤1.5 x Upper Limit Normal (ULN). NB: This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
11. Adequate liver function:

    * Total bilirubin ≤1.5 X ULN (<3.0 x ULN for patients with Gilbert's syndrome)
    * Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≤2.5 x ULN
12. Adequate renal function: Measured creatinine clearance ≥40 mL/min or calculated creatinine clearance ≥40 mL/min using Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
13. Life expectancy of ≥6 months
14. Willing and able to give informed consent (which includes compliance with the requirements and restrictions listed in the patient information sheet (PIS) and in this protocol). NB: Consent must be obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
15. Patients of child-bearing potential and male patients with female partners of child-bearing potential must agree to use highly effective contraception methods from date of consent, which must be continued for up to 90 days after last treatment administration.
16. Female patients must not be pregnant. There should be sufficient evidence of post-menopausal status or a negative serum pregnancy test for pre-menopausal female patients.
17. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and any other study procedures.

Exclusion Criteria:

1. Any history of autoimmune or inflammatory disease including (any patients with a history of an autoimmune condition but without active disease in the last 5 years may be included only after consultation with the CI/TMG):

   * Inflammatory bowel disease (e.g. colitis or Crohn's disease)
   * Diverticulitis (with the exception of diverticulosis)
   * Systemic lupus erythematous (SLE)
   * Sarcoidosis syndrome
   * Wegener syndrome (granulomatosis with polyangitis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis, etc.)
2. Patients with prior allogeneic stem cell or solid organ transplantation
3. Patients who have had prior treatment with anti- PD-1, PD-L1 or CTLA-4 monoclonal antibody or other novel immune-oncology agent(s)
4. Active invasive malignancy in the previous 2 years excluding non-melanoma skin cancer
5. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia) or evidence of active pneumonitis on screening chest CT scan (history of radiation pneumonitis in the radiation field is permitted)
6. Patients with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
7. QTcF value of >470 ms. If prolonged, this should be confirmed by 2 further ECGs each separated by at least 5 minutes.
8. Patients with the following risk factors for bowel perforation:

   * History of acute diverticulitis or intra-abdominal abcess in the last 3 years
   * History of mechanical GI obstruction or abdominal carcinomatosis
9. Any unresolved toxicity CTCAE Grade ≥2 from previous anti-cancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Patients with any irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the CI/TMG
10. Receipt of last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, embolisation, monoclonal antibodies) within 30 days prior to first dose of trial treatment. NB: If sufficient washout time has not occurred due to the schedule or pharmacokinetic (PK) properties of an agent, a longer washout period will be required, as agreed by the Trial Management Group (TMG) and/or Chief Investigator (CI).
11. Treatment with any experimental drug within 30 days or 5 half-lives (whichever is longer) of the first dose of trial treatment
12. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
13. Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial
14. Received therapeutic oral antibiotics that cannot be discontinued at least 14 days prior to starting treatment or received intravenous (IV) antibiotics within 14 days prior to registration. NB: Patients receiving prophylactic antibiotics (e.g. for prevention of a urinary tract infection or COPD) are eligible
15. Any psychiatric or other disorder (e.g. brain metastases) that impacts the patients ability to give informed consent or comply with trial treatment and activities
16. History of leptomeningeal carcinomatosis
17. Active infection of tuberculosis (TB) (clinically evaluated in accordance with local guidelines, e.g. clinical history, examination and radiographic findings with or without TB testing as clinically indicated)
18. Patients must not have had systemic corticosteroid therapy (>10 mg daily prednisolone equivalent) within 14 days prior to registration or concomitant use of other immunosuppressive medications. NB: The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e. for adrenal insufficiency) and mineralocorticoids (e.g. fludrocortisone) are allowed
19. Administration of a live, attenuated vaccine within 4 weeks prior to planned start of treatment or anticipation that such a live, attenuated vaccine will be required during the study
20. Evidence of significant uncontrolled concomitant disease that could substantially increase the risk of incurring adverse events (AEs), affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis), uncontrolled hypertension, serious chronic gastrointestinal conditions associated with diarrhoea and uncontrolled major seizure disorder
21. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of trial treatment. This does not include rigid cystoscopy and biopsies
22. Significant cardiovascular disease, such as:

    * New York Heart Association cardiac disease (Class II or greater)
    * Myocardial infarction within 3 months prior to registration
    * Unstable arrhythmias
    * Unstable angina
23. Patients with uncontrolled Type 1 diabetes mellitus. Patients controlled on a stable insulin regimen are eligible
24. Patients with uncontrolled adrenal insufficiency
25. Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
26. Known active primary immune deficiency, including but not limited to, uncontrolled human immunodeficiency virus (HIV) (detectable viral load) or acquired immunodeficiency syndrome (AIDS)-related illness
27. Women who are pregnant or breast feeding. Female or male patient of reproductive potential who is not willing to employ highly effective birth control from screening to 90 days after the last dose of trial treatment.
28. Known allergy or hypersensitivity to any of the investigational products or their excipients
29. Prior enrolment to, or treatment in a previous durvalumab clinical study, regardless of treatment arm assignment
30. Patients must not donate blood while participating in this study and for at least 90 days following the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity (Phase 1b) | At the end of cycle 1 (cycle 1 is 28 days)
  Detailed adverse event monitoring will be conducted, assessed using CTCAE v5. Dose Limiting Toxicity (DLT) is defined as any adverse event or laboratory abnormality detailed in the trial protocol, that has a reasonable possibility of being related to trial treatment and occurring at anytime during the DLT evaluation period (28 days from the first administration of S-488210/S-488211 on cycle 1 day 2).
Pathological Disease Free Survival Rate (DFSR) (Phase 2) | 1 year after start of treatment
  Disease Free Survival will be calculated from start of trial treatment (cycle 1 day 1) until the time at which either primary disease is confirmed to have recurred, any secondary cancer is confirmed or death from any cause. The primary endpoint of Disease Free Survival Rate will be assessed at 1 year from start of treatment (and include patients that start trial treatment and receive combination treatment on cycle 2 day 1) and compared to the historical control rate of 20%.

SECONDARY OUTCOMES:
1 year DFSR stratified by HLA-A*02:01 | 1 year after start of treatment
  If the primary endpoint (DFSR) is statistically signification, comparison of DFSR at 1 year will be conducted between patients that are human leukocyte antigen-A (HLA-A*02:01) positive versus negative.
5 year Overall Survival rate | 5 years from start of treatment to date of death, if applicable.
  Overall survival will be assessed from time of starting treatment to time of death from any cause.
5 year Overall Survival rate stratified by HLA-A*02:01 | 5 years from start of treatment to date of death, if applicable.
  Overall survival will be assessed from time of starting treatment to time of death from any cause, stratified by HLA-A*02:01 positive or negative.
Assessment of Quality of Life using EORTC QLQ-C30 questionnaire | Assessments will be performed at baseline (prior to starting treatment on cycle 1 days 1), every 12 weeks up to 12 months after start of treatment and 24 months after start of treatment.
  Quality of Life assessments will be undertaken using EORTC QLQ-C30 (version 3) questionnaire using Likert score (26 questions scored: 1=not at all, 2=a little, 3=quite a bit, 4=very much; 2 questions scored: 1-7, 1=very poor, 7=excellent) . Descriptions of mean change in EORTC QLQ scores will be presented and compared to baseline values from pre-treatment.
Assessment of Quality of Life using EORTC QLQ-NMIBC24 questions | Assessments will be performed at baseline (prior to starting treatment on cycle 1 days 1), every 12 weeks up to 12 months after start of treatment and 24 months after start of treatment.
  Quality of Life assessments will be undertaken using EORTC QLQ-C30 which will include QLQ-NMIBC24 questions using Likert score (24 questions scored: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Descriptions of mean change in EORTC QLQ scores will be presented and compared to baseline values from pre-treatment.
Assessment of Quality of Life using EQ-5D-5L questionnaire | Assessments will be performed at baseline (prior to starting treatment on cycle 1 days 1), every 12 weeks up to 12 months after start of treatment and 24 months after start of treatment.
  Quality of Life assessments will be undertaken using EQ-5D-5L (self-reported) questionnaire using a combination of Likert score (5 questions with 5 dimensions of abilities) and visual analogue score (scored 0-100, 0=worst, 100=best). Descriptions of mean change in EQ-5D-5L scores will be presented and compared to baseline values from pre-treatment.

OTHER OUTCOMES:
1 year DFSR stratified by PD-L1 status | 1 year after start of treatment
  DFSR at 1 year stratified, retrospectively, by PD-L1 status will be performed.
1 year DFSR stratified by baseline Tumour Infiltrating Lymphocyte (TIL) status | 1 year after start of treatment
  DFSR at 1 year stratified, retrospectively, by TIL status (high, intermediate and low) to assess the distribution of a three-category variable (TIL status) over survival status.
5 year Overall Survival rate stratified by PD-L1 status and TIL status | 5 years from start of treatment to date of death, if applicable.
  Overall survival will be assessed from time of starting treatment to time of death from any cause, stratified by PD-L1 status and TIL status.
Correlation of plasma cytokine levels with 1 year DFSR | 1 year after start of treatment
  The association between DFSR at 1 year and plasma cytokine levels will be assessed using logistic regression, with odds ratios and 95% confidence interval reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Linch, Principal Investigator — University College London Hospital
Locations (5):
- United Kingdom (5):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No